CLINICAL TRIAL: NCT05896748
Title: An Amendment to the FLAIR Study to Evaluate the Pharmacokinetics, Safety, Tolerability, Maintenance of Virological Suppression and Patient Reported Outcomes for Participants Receiving Cabotegravir (CAB 200 mg/mL) and Rilpivirine (300 mg/mL) Long-Acting Injections Following Sub-cutaneous (SC) Administration in the Anterior Abdominal Wall SC Tissue Compared With Intramuscular (IM) Administration in the Gluteus Medius Muscle in Adult Participants Living With HIV-1 Infection in the FLAIR Study
Brief Title: Study to Assess the Effects of Cabotegravir (CAB) and Rilpivirine (RPV) Long-Acting (LA) Injections Following Sub-cutaneous (SC) Administration Compared With Intramuscular (IM) Administration in Adult Participants Living With Human Immunodeficiency Virus (HIV-1) Infection in the FLAIR Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201584-001
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1)
Keywords: Antiretroviral agent; Rilpivirine; Cabotegravir; FLAIR; Human immunodeficiency virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg (Experimental): Participants received an intramuscular (IM) injection of CAB LA 400 mg and RPV LA 600 mg on week -4 during the Screening phase. Participants then received a sub-cutaneous (SC) injection of CAB LA 400 mg + RPV LA 600 mg on Day 1 of Week 1, Week 4 and Week 8 (once in every 4 weeks (Q4W)) for a total of 12 weeks during the SC abdominal Injection Phase. 4 weeks later, participants returned to the clinic for an IM gluteal injection (at Week 12) of CAB LA 400 mg + RPV LA 600 mg during the Return to Gluteal Injection Phase and subsequent gluteal injection occurred after Q4W at Week 16.
  Interventions: Drug: Cabotegravir - Injectable Suspension (CAB LA); Drug: Rilpivirine - Injectable Suspension (RPV LA)

INTERVENTIONS:
Drug: Cabotegravir - Injectable Suspension (CAB LA) — It is a sterile white to slightly pink suspension containing 200 mg/mL of CAB as free acid for administration by intramuscular (IM) injection. Each vial is for single-dose use containing a withdrawable volume of 2.0 mL, and does not require dilution prior to administration. CAB LA is composed of cabotegravir free acid, polysorbate 20, polyethylene glycol 3350, mannitol, and water for injection.
Drug: Rilpivirine - Injectable Suspension (RPV LA) — It is a sterile white suspension containing 300 mg/mL of RPV as the free base. The route of administration is by intramuscular (IM) injection. Each vial contains a nominal fill of 2.0 mL, and does not require dilution prior to administration. RPV LA requires refrigeration and must be protected from light. RPV LA is composed of RPV free base, poloxamer 338, sodium dihydrogen phosphate monohydrate, citric acid monohydrate, glucose monohydrate, sodium hydroxide, water for injection.

SUMMARY:
This study will assess the pharmacokinetics, safety, tolerability, maintenance of virological suppression and patient reported outcomes for participants receiving CAB and RPV LA injections following SC administration in the anterior abdominal wall SC tissue compared with IM administration in the gluteus medius muscle in adult participants living with HIV-1 infection in the FLAIR study (NCT02938520).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent (FLAIR and Sub-study specific informed consent)
* Eligible participants must have been on CAB LA + RPV LA regimen for a minimum of 12 months while on the FLAIR study. Any disruptions in dosing during FLAIR must be discussed with the Medical Monitor for a final determination of eligibility into the sub-study.
* Plasma HIV-1 RNA <50 c/mL at Sub-Study Screening.
* History of Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) vaccination (or booster dosing) is allowed prior to sub study screening and will be allowed during the conduct of the sub-study as long as the vaccine (or boosters) are not administered within 14 days of virologic load (VL) assessments.
* HIV-1 infected antiretroviral therapy (ART)-naive men or women aged 18 years or greater at the time of signing the informed consent.
* HIV-1 infection as documented by Screening plasma HIV-1 RNA >=1000 cubic (c)/mL
* Antiretroviral-naive (less than or equal to (<=10) days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection). Any previous exposure to an HIV integrase inhibitor or non-nucleoside reverse transcriptase inhibitor will be exclusionary
* Female Participants: A female participant is eligible to participate if she is not pregnant at Screening and first day of Induction Phase (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies

  1. Non-reproductive potential defined as:

     * Pre-menopausal females with one of the following:
     * Documented tubal ligation;
     * Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion;
     * Hysterectomy; Documented Bilateral Oophorectomy;
     * Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.
  2. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, and for at least 30 days after discontinuation of all oral study medications and for at least 52 weeks after discontinuation of CAB LA and RPV LA.
* The investigator is responsible for ensuring that participants understand how to properly use these methods of contraception.
* All participants in the study should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (example [e.g.,] male condom) and on the risk of HIV transmission to an uninfected partner.
* In France, a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* More than 1 plasma HIV-1 RNA measurement 50 c/mL to <200 c/mL (virologic blip) within 24 weeks prior to sub-study Screening visit that was investigated and found NOT to be associated with alternative causes including recent vaccinations received within 4 weeks of the viral blip or NOT associated with intercurrent illness that developed within 2-4 weeks of the viral blip.
* All viral blips that occurred within 24 weeks prior to screening should be discussed with the Medical Monitor to assess whether such a participant can enroll into the sub-study.
* Any Suspected Virologic Failure (HIV-RNA 200 c/mL) as defined during FLAIR study.
* Participants planning to require oral bridging during participation in the FLAIR sub study.
* The participant has a tattoo or any dermatological condition overlying the abdominal or gluteal regions which may interfere with interpretation of injection site reactions.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* Any woman of childbearing potential who is pregnant at screening will be excluded from entering the sub-study.
* Any women of childbearing potential who gets pregnant while on the sub-study will have to be withdrawn from the sub-study but will be allowed to transition back to the parent FLAIR study if a pregnancy specific Informed Consent Form (ICF) is signed, and commercial access is not available at the time of pregnancy
* Women who are pregnant, breastfeeding, or plan to become pregnant or breastfeed during the study.
* Any evidence at Screening of an active Centers for Disease and Prevention Control (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy or historic or current cluster of differentiation 4+ (CD4+) cell count <200 cells/ cubic millimeter (mm^3) are not exclusionary.
* Participants with known moderate to severe hepatic impairment.
* Any pre-existing physical or mental condition (including substance abuse disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrollment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrollment.
* Participant who, in the investigator's judgment, poses a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* The participant has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti HBc), Hepatitis B surface antibody (anti-HBs) and HBV Deoxyribonucleic acid (DNA) as follows:

  * Participants positive for HBsAg are excluded;
  * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.
* Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; participants who are anticipated to require HCV treatment prior to Week 48 of the Maintenance Phase must be excluded. HCV treatment on study may be permitted post Week 48, following consultation with the Medical Monitor. Participants with HCV co-infection will be allowed entry into Phase 3 studies if:

  * Liver enzymes meet entry criteria;
  * HCV Disease has undergone appropriate work-up, HCV is not advanced, and will not require treatment prior to the Week 48 visit. Additional information (where available) on participants with HCV co-infection at screening should include results from any liver biopsy, fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment.
  * In the event that recent biopsy or imaging data is not available or is inconclusive, the Fib-4 score will be used to verify eligibility.
  * A Fib-4 score > 3.25 is exclusionary;
  * Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation. Fibrosis 4 Score Formula: (Age * AST)/ (Platelets * [square root of ALT]).
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis.
* All participants will be screened for syphilis (rapid plasma reagin [RPR]). Participants with untreated syphilis infection, defined as a positive RPR without clear documentation of treatment, are excluded. Participants with a positive RPR test who have not been treated may be rescreened at least 30 days after completion of antibiotic treatment for syphilis.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the study Medical Monitor for inclusion of the participant prior to enrollment.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the drug or render the participant unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during pharmacokinetic (PK) sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.
* Current or anticipated need for chronic anti-coagulation.
* ALT >=3 times upper limit normal (ULN).
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Exposure to an experimental drug and/or experimental vaccine within 28 days or 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product (IP).
* Treatment with any of the following agents within 28 days of Screening:

  * radiation therapy;
  * cytotoxic chemotherapeutic agents;
  * tuberculosis (TB) therapy, with the exception of treatment of latent TB with isoniazid;
  * Immunomodulators that alter immune responses (such as chronic systemic corticosteroids, interleukins, or interferons).
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 within 28 days of the first dose of IP.
* Use of medications which are associated with Torsades de Pointes
* Any evidence of primary resistance to non-nuclease reverse transcriptase inhibitors (NNRTIs) (except for K103N which is allowed), or any known resistance to Integrase inhibitors from historical resistance test results.
* Participants who are human leukocyte antigen (HLA)-B*5701 positive and are unable to use an NRTI backbone that does not contain abacavir (participants who are HLA-B*5701 positive may be enrolled if they use a nuclease reverse transcriptase inhibitors (NRTI) backbone that does not contain abacavir; HLA-B*5701 positive participants may be excluded from the study if local provision of an alternate NRTI backbone is not possible).
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening Phase to verify a result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the participant's participation in the study of an investigational compound.
* Participant has estimated creatinine clearance <50 mL/minute (min)/1.73 meter square (m^2) via the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Participants who are currently participating in or anticipate to be selected for any other interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (26):
- United States (5):
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
- GSK Investigational Site, Toronto, Ontario, Canada
- Japan (2):
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- South Africa (3):
  - GSK Investigational Site, Bloemfontein, Free State
  - GSK Investigational Site, Wentworth, KwaZulu-Natal
  - GSK Investigational Site, Durban
- Spain (12):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Ferrol
  - GSK Investigational Site, Granada
  - GSK Investigational Site, La Laguna-Tenerife
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, San Sebastián de los Reyes
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Santander
- United Kingdom (3):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The sub-study Safety population, which included all enrolled participants who received at least 1 subcutaneous (SC) injection, was used to present the baseline characteristics and outcome measures.
  Participant flow was presented for the overall group, adverse events were presented phase wise and outcome measures were presented for the overall group or treatment wise (per dose or per overall treatment received).
Period: Screening Phase (Week -4 up to Day 1)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Started | 94
Completed | 93
Not Completed | 1
Not completed — Passed away due to unknown reasons | 1
Period: SC Injection Phase (Day 1 up to Week 12)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Started | 93
Completed | 87
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3
Period: Return to IM Glu Inj Phase(Week12-Week20
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Started | 87
Completed | 86
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics presented based on sub-study Safety population. Summary of baseline/demographics for some race/ ethnicity variables are presented as de-identified to prevent risk of participant re-identification.
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 19
  White - White/Caucasian/European Heritage | 63
  De-identified | 11

OUTCOME MEASURES:

1. Primary Outcome: Concentrations at the End of the Dosing Interval (Ctau) of CAB LA 400 mg Following Administration CAB LA + RPV LA
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: At screening Week-4; Day 1, Week 4, Week 8 for SC injections; and Week 12 for Return to IM gluteal injection
Population: Analysis was performed on sub-study Pharmacokinetic (PK) parameter set for CAB LA, which included all participants who received at least one CAB and/or RPV SC injection and had evaluable Ctau parameter estimated during the sub-study period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- CAB+RPV Screening Gluteal Injection: Participants received an IM gluteal injections of CAB LA 400 mg and RPV LA 600 mg at Week -4 during Screening/IM Gluteal Injection Phase.
- CAB+RPV First Sub-Cutaneous (SC) Injection: Participants received a first SC injection of CAB LA 400 mg and RPV LA 600 mg on Day 1 during SC abdominal injection phase.
- CAB+RPV Second SC Injection: Participants received a second SC injection of CAB LA 400 mg and RPV LA 600 mg on Week 4 during SC abdominal injection phase.
- CAB+RPV Last SC Injection: Participants received a last SC injection of CAB LA 400 mg and RPV LA 600 mg on Week 8 during SC abdominal injection phase.
- CAB+RPV Return to Intramuscular (IM) Gluteal Injection: Participants received an IM gluteal injection of CAB LA 400 mg and RPV LA 600 mg on Week 12 and Week 16 during Return to IM gluteal injection phase
Arm/Group | CAB+RPV Screening Gluteal Injection | CAB+RPV First Sub-Cutaneous (SC) Injection | CAB+RPV Second SC Injection | CAB+RPV Last SC Injection | CAB+RPV Return to Intramuscular (IM) Gluteal Injection
Number analyzed (Participants) | 81 | 74 | 84 | 78 | 85
microgram per milliliter (µg/mL) | 2.759 (36.64) | 2.670 (37.02) | 2.607 (39.00) | 2.632 (38.87) | 2.797 (36.18)
Statistical Analysis 1: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV First Sub-Cutaneous (SC) Injection; To compare the abdominal SC injection with gluteal IM injection for Ctau within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.948, 90% CI 2-sided [0.901 to 0.998]
Statistical Analysis 2: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Second SC Injection; To compare the abdominal SC injection with gluteal IM injection for Ctau within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.935, 90% CI 2-sided [0.877 to 0.995]
Statistical Analysis 3: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Last SC Injection; To compare the abdominal SC injection with gluteal IM injection for Ctau within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.934, 90% CI 2-sided [0.872 to 1.000]
Statistical Analysis 4: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Return to Intramuscular (IM) Gluteal Injection; To compare the IM gluteal injections for Ctau within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.999, 90% CI 2-sided [0.943 to 1.059]

2. Primary Outcome: Ctau of RPV LA 600 mg Following Administration of CAB LA + RPV LA
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: At screening Week-4; Day 1, Week 4, Week 8 for SC abdominal injections; and Week 12 for Return to IM gluteal injection
Population: Analysis was performed on sub-study PK parameter set for RPV LA, which included all participants who received at least one CAB and/or RPV SC injection and had evaluable Ctau parameter estimated during the sub-study period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | CAB+RPV Screening Gluteal Injection | CAB+RPV First Sub-Cutaneous (SC) Injection | CAB+RPV Second SC Injection | CAB+RPV Last SC Injection | CAB+RPV Return to Intramuscular (IM) Gluteal Injection
Number analyzed (Participants) | 80 | 75 | 84 | 77 | 84
Nanograms per milliliter (ng/mL) | 137.021 (38.51) | 138.611 (36.43) | 135.620 (35.55) | 128.590 (39.71) | 139.879 (43.06)
Statistical Analysis 1: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV First Sub-Cutaneous (SC) Injection; To compare the abdominal SC injection with gluteal IM injection for Ctau within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 1.002, 90% CI 2-sided [0.952 to 1.056]
Statistical Analysis 2: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Second SC Injection; To compare the abdominal SC injection with gluteal IM injection for Ctau within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.961, 90% CI 2-sided [0.921 to 1.002]
Statistical Analysis 3: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Last SC Injection; To compare the abdominal SC injection with gluteal IM injection for Ctau within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.928, 90% CI 2-sided [0.885 to 0.973]
Statistical Analysis 4: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Return to Intramuscular (IM) Gluteal Injection; To compare the IM gluteal injections for Ctau within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 1.003, 90% CI 2-sided [0.955 to 1.053]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) One Week Post Dose of CAB LA 400 mg Following Administration of CAB LA + RPV LA
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: At screening week -3; Week 1, Week 5, Week 9 for SC abdominal injections; and Week 13 for Return to IM gluteal injection
Population: Analysis was performed on sub-study PK parameter set for CAB LA, which included all participants who received at least one CAB and/or RPV SC injection and had evaluable Cmax parameter estimated during the sub-study period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | CAB+RPV Screening Gluteal Injection | CAB+RPV First Sub-Cutaneous (SC) Injection | CAB+RPV Second SC Injection | CAB+RPV Last SC Injection | CAB+RPV Return to Intramuscular (IM) Gluteal Injection
Number analyzed (Participants) | 90 | 92 | 89 | 86 | 85
µg/mL | 3.545 (34.77) | 3.316 (35.22) | 3.165 (36.77) | 3.215 (34.56) | 3.529 (37.05)
Statistical Analysis 1: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV First Sub-Cutaneous (SC) Injection; To compare the abdominal SC injection with gluteal IM injection for Cmax within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.942, 90% CI 2-sided [0.897 to 0.990]
Statistical Analysis 2: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Second SC Injection; To compare the abdominal SC injection with gluteal IM injection for Cmax within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.911, 90% CI 2-sided [0.860 to 0.965]
Statistical Analysis 3: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Last SC Injection; To compare the abdominal SC injection with gluteal IM injection for Cmax within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.910, 90% CI 2-sided [0.857 to 0.966]
Statistical Analysis 4: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Return to Intramuscular (IM) Gluteal Injection; To compare the IM gluteal injections for Cmax within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 1.003, 90% CI 2-sided [0.938 to 1.074]

4. Primary Outcome: Cmax One Week Post Dose of RPV LA 600 mg Following Administration of CAB LA + RPV LA
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: as for outcome 3
Population: Analysis was performed on sub-study PK parameter set for RPV LA, which included all participants who received at least one CAB and/or RPV SC injection and had evaluable Cmax parameter estimated during the sub-study period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CAB+RPV Screening Gluteal Injection | CAB+RPV First Sub-Cutaneous (SC) Injection | CAB+RPV Second SC Injection | CAB+RPV Last SC Injection | CAB+RPV Return to Intramuscular (IM) Gluteal Injection
Number analyzed (Participants) | 89 | 92 | 89 | 86 | 84
ng/mL | 162.287 (35.73) | 152.614 (36.56) | 148.051 (35.27) | 149.145 (36.91) | 154.659 (36.38)
Statistical Analysis 1: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV First Sub-Cutaneous (SC) Injection; To compare the abdominal SC injection with gluteal IM injection for Cmax within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.938, 90% CI 2-sided [0.895 to 0.982]
Statistical Analysis 2: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Second SC Injection; To compare the abdominal SC injection with gluteal IM injection for Cmax within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.918, 90% CI 2-sided [0.876 to 0.963]
Statistical Analysis 3: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Last SC Injection; To compare the abdominal SC injection with gluteal IM injection for Cmax within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.905, 90% CI 2-sided [0.861 to 0.952]
Statistical Analysis 4: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Return to Intramuscular (IM) Gluteal Injection; To compare the IM gluteal injections for Cmax within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.937, 90% CI 2-sided [0.891 to 0.986]

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 Through the End of Dosing Interval (AUC[0-tau]) of CAB LA 400 mg Following Administration of CAB LA + RPV LA
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: At screening Week-4; Day 1, Week 4, Week 8 for SC abdominal injections; and Week 12, for Return to IM gluteal injection
Population: Analysis was performed on sub-study PK parameter set for CAB LA, which included all participants who received at least one CAB and/or RPV SC injection and had evaluable AUC[0-tau] parameter estimated during the sub-study period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour microgram per milliliter (h*µg/mL)
Arm/Group | CAB+RPV Screening Gluteal Injection | CAB+RPV First Sub-Cutaneous (SC) Injection | CAB+RPV Second SC Injection | CAB+RPV Last SC Injection | CAB+RPV Return to Intramuscular (IM) Gluteal Injection
Number analyzed (Participants) | 80 | 73 | 82 | 78 | 85
hour microgram per milliliter (h*µg/mL) | 2051.172 (34.31) | 1997.801 (33.94) | 1943.596 (35.25) | 1943.787 (35.53) | 2155.520 (32.71)
Statistical Analysis 1: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV First Sub-Cutaneous (SC) Injection; To compare the abdominal SC injection with gluteal IM injection for AUC[0-tau] within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.944, 90% CI 2-sided [0.906 to 0.983]
Statistical Analysis 2: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Second SC Injection; To compare the abdominal SC injection with gluteal IM injection for AUC[0-tau] within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.944, 90% CI 2-sided [0.895 to 0.995]
Statistical Analysis 3: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Last SC Injection; To compare the abdominal SC injection with gluteal IM injection for AUC[0-tau] within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.933, 90% CI 2-sided [0.876 to 0.994]
Statistical Analysis 4: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Return to Intramuscular (IM) Gluteal Injection; To compare the IM gluteal injections for AUC[0-tau] within CAB; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 1.040, 90% CI 2-sided [0.979 to 1.105]

6. Primary Outcome: AUC[0-tau] of RPV LA 600 mg Following Administration of CAB LA + RPV LA
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: At screening Week-4; Day 1, Week 4, Week 8 for SC abdominal injections; and Week 12 for Return to IM gluteal injection
Population: Analysis was performed on sub-study PK parameter set for RPV LA, which included all participants who received at least one CAB and/or RPV SC injection and had evaluable AUC[0-tau] parameter estimated during the sub-study period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | CAB+RPV Screening Gluteal Injection | CAB+RPV First Sub-Cutaneous (SC) Injection | CAB+RPV Second SC Injection | CAB+RPV Last SC Injection | CAB+RPV Return to Intramuscular (IM) Gluteal Injection
Number analyzed (Participants) | 78 | 73 | 83 | 77 | 83
h*µg/mL | 98003.488 (34.31) | 98801.696 (35.32) | 95743.414 (34.56) | 93248.069 (34.85) | 100006.767 (34.78)
Statistical Analysis 1: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV First Sub-Cutaneous (SC) Injection; To compare the abdominal SC injection with gluteal IM injection for AUC[0-tau] within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.966, 90% CI 2-sided [0.932 to 1.002]
Statistical Analysis 2: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Second SC Injection; To compare the abdominal SC injection with gluteal IM injection for AUC[0-tau] within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.955, 90% CI 2-sided [0.922 to 0.989]
Statistical Analysis 3: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Last SC Injection; To compare the abdominal SC injection with gluteal IM injection for AUC[0-tau] within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 0.948, 90% CI 2-sided [0.907 to 0.991]
Statistical Analysis 4: Comparison: CAB+RPV Screening Gluteal Injection vs CAB+RPV Return to Intramuscular (IM) Gluteal Injection; To compare the IM gluteal injections for AUC[0-tau] within RPV; Test type: Other; Mixed effect analysisofcovariance(ANCOVA; Ratio of geometric least square mean = 1.014, 90% CI 2-sided [0.972 to 1.058]

7. Secondary Outcome: Number of Participants With Injection Site Reactions (ISRs) and by Maximum Severity - SC Injection Phase
Description: Severity of ISRs was analyzed using division of acquired immunodeficiency syndrome (DAIDS) grading scale. The severity is categorized into grades as following: Grade 1 - mild, Grade 2 - moderate, Grade 3 - severe, Grade 4 - Potentially life threatening, Grade 5 - Death. Higher grade indicates more severe condition.
Time Frame: From Day 1 Up to Week 12
Population: Analysis was performed on sub-study safety set, which included all enrolled participants who received at least one CAB and/or RPV SC injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Participants
  ISRs | 85
  Mild or Grade 1 ISRs | 43
  Moderate or Grade 2 ISRs | 36
  Severe or Grade 3 ISRs | 6
  Potentially Life-Threatening or Grade 4 ISRs | 0
  Death or Grade 5 ISRs | 0

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) Based on Maximum Severity Grade - SC Injection Phase
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Severity of AESI was analyzed using DAIDS grading scale. The severity is categorized into grades as following: Grade 1 - mild, Grade 2 - moderate, Grade 3 - severe, Grade 4 - Potentially life threatening, Grade 5 - Death. Higher grade indicates more severe condition. AESI assessed were Depression, Anxiety, Impact on creatinine, Hyperglycaemia.
Time Frame: From Day 1 Up to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Participants
  Any Depression | 1
  Mild or Grade 1 Depression | 0
  Moderate or Grade 2 Depression | 1
  Severe or Grade 3 Depression | 0
  Potentially Life-Threatening or Grade 4 Depression | 0
  Death or Grade 5 Depression | 0
  Any Anxiety | 1
  Mild or Grade 1 Anxiety | 1
  Moderate or Grade 2 Anxiety | 0
  Severe or Grade 3 Anxiety | 0
  Potentially Life-Threatening or Grade 4 Anxiety | 0
  Death or Grade 5 Anxiety | 0
  Any Impact on Creatinine | 1
  Mild or Grade 1 Impact on Creatinine | 1
  Moderate or Grade 2 Impact on Creatinine | 0
  Severe or Grade 3 Impact on Creatinine | 0
  Potentially Life-Threatening or Grade 4 Impact on Creatinine | 0
  Death or Grade 5 Impact on Creatinine | 0
  Any Hyperglycaemia | 1
  Mild or Grade 1 Hyperglycaemia | 1
  Moderate or Grade 2 Hyperglycaemia | 0
  Severe or Grade 3 Hyperglycaemia | 0
  Potentially Life-Threatening or Grade 4 Hyperglycaemia | 0
  Death or Grade 5 Hyperglycaemia | 0

9. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to ISRs and AESIs - SC Injection Phase
Time Frame: From Day 1 Up to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Participants
  Discontinuations due to ISR | 5
  Discontinuations due to AESI | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) From the Last IM Gluteal Injection in Screening Phase to the End of the SC Injection Phase
Description: SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs.
Time Frame: From Week -4 Up to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Participants
  Any AEs | 90
  Any SAEs | 0

11. Secondary Outcome: Change From Baseline in Chemistry Parameters Following Administration of SC Injection: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), and Creatine Phosphokinase
Description: Blood samples were collected as assessed by protocol, at specific time points for the analysis of clinical chemistry parameters. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: Analysis was performed on sub-study safety set, which included all enrolled participants who received at least one CAB and/or RPV SC injection. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
International units per liter (IU/L)
  ALT, Baseline (screening Week -4) | 21.6 (10.38)
  ALT, CFB at Week 4: number analyzed (Participants) | 90
  ALT, CFB at Week 4 | 1.2 (8.09)
  ALT, CFB at Week 8: number analyzed (Participants) | 85
  ALT, CFB at Week 8 | -0.4 (5.94)
  ALT, CFB at Week 12: number analyzed (Participants) | 86
  ALT, CFB at Week 12 | -0.7 (7.32)
  ALP, Baseline (screening Week -4) | 62.3 (14.72)
  ALP, CFB at Week 4: number analyzed (Participants) | 90
  ALP, CFB at Week 4 | -0.1 (7.51)
  ALP, CFB at Week 8: number analyzed (Participants) | 85
  ALP, CFB at Week 8 | 0.7 (6.66)
  ALP, CFB at Week 12: number analyzed (Participants) | 86
  ALP, CFB at Week 12 | -0.4 (6.29)
  AST, Baseline (screening Week -4) | 20.1 (6.27)
  AST, CFB at Week 4: number analyzed (Participants) | 90
  AST, CFB at Week 4 | 2.2 (12.33)
  AST, CFB at Week 8: number analyzed (Participants) | 85
  AST, CFB at Week 8 | 0.1 (5.52)
  AST, CFB at Week 12: number analyzed (Participants) | 86
  AST, CFB at Week 12 | -0.2 (5.46)
  Creatine phosphokinase, Baseline (screening Week -4) | 166.8 (163.38)
  Creatine phosphokinase, CFB at Week 4: number analyzed (Participants) | 90
  Creatine phosphokinase, CFB at Week 4 | 47.7 (340.57)
  Creatine phosphokinase, CFB at Week 8: number analyzed (Participants) | 85
  Creatine phosphokinase, CFB at Week 8 | 3.3 (206.30)
  Creatine phosphokinase, CFB at Week 12: number analyzed (Participants) | 86
  Creatine phosphokinase, CFB at Week 12 | -0.9 (162.90)

12. Secondary Outcome: Change From Baseline in Chemistry Parameters Following Administration of SC Injection: Creatinine, Total Bilirubin
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Micromoles per liter (umol/L)
  Creatinine, Baseline (screening Week -4) | 86.23 (14.551)
  Creatinine, CFB at Week 4: number analyzed (Participants) | 90
  Creatinine, CFB at Week 4 | -1.84 (5.811)
  Creatinine, CFB at Week 8: number analyzed (Participants) | 85
  Creatinine, CFB at Week 8 | -1.55 (8.224)
  Creatinine, CFB at Week 12: number analyzed (Participants) | 86
  Creatinine, CFB at Week 12 | -0.35 (7.206)
  Total Bilirubin, Baseline (screening Week -4) | 9.2 (4.01)
  Total Bilirubin, CFB at Week 4: number analyzed (Participants) | 90
  Total Bilirubin, CFB at Week 4 | 0.5 (3.52)
  Total Bilirubin, CFB at Week 8: number analyzed (Participants) | 85
  Total Bilirubin, CFB at Week 8 | -0.5 (3.64)
  Total Bilirubin, CFB at Week 12: number analyzed (Participants) | 86
  Total Bilirubin, CFB at Week 12 | -1.2 (3.21)

13. Secondary Outcome: Change From Baseline in Chemistry Parameters Following Administration of SC Injection: Glucose, Potassium, Sodium, Blood Urea Nitrogen, Carbon Dioxide, Chloride, Phosphate
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Millimoles per liter (mmol/L)
  Glucose, Baseline (screening Week -4): number analyzed (Participants) | 89
  Glucose, Baseline (screening Week -4) | 5.14 (0.808)
  Glucose, CFB at Week 12: number analyzed (Participants) | 85
  Glucose, CFB at Week 12 | -0.02 (0.571)
  Potassium, Baseline (screening Week -4) | 4.19 (0.304)
  Potassium, CFB at Week 4: number analyzed (Participants) | 90
  Potassium, CFB at Week 4 | 0.02 (0.389)
  Potassium, CFB at Week 8: number analyzed (Participants) | 85
  Potassium, CFB at Week 8 | 0.03 (0.307)
  Potassium, CFB at Week 12: number analyzed (Participants) | 86
  Potassium, CFB at Week 12 | -0.04 (0.346)
  Sodium, Baseline (screening Week -4) | 139.8 (1.81)
  Sodium, CFB at Week 4: number analyzed (Participants) | 90
  Sodium, CFB at Week 4 | -0.1 (1.72)
  Sodium, CFB at Week 8: number analyzed (Participants) | 85
  Sodium, CFB at Week 8 | 0.4 (2.11)
  Sodium, CFB at Week 12: number analyzed (Participants) | 86
  Sodium, CFB at Week 12 | 0.3 (1.91)
  Blood Urea Nitrogen, Baseline (screening Week -4) | 5.33 (1.639)
  Blood Urea Nitrogen, CFB at Week 4: number analyzed (Participants) | 90
  Blood Urea Nitrogen, CFB at Week 4 | 0.13 (1.206)
  Blood Urea Nitrogen, CFB at Week 8: number analyzed (Participants) | 85
  Blood Urea Nitrogen, CFB at Week 8 | 0.22 (1.417)
  Blood Urea Nitrogen, CFB at Week 12: number analyzed (Participants) | 86
  Blood Urea Nitrogen, CFB at Week 12 | -0.04 (1.368)
  Carbon Dioxide, Baseline (screening Week -4) | 23.6 (2.04)
  Carbon Dioxide, CFB at Week 4: number analyzed (Participants) | 90
  Carbon Dioxide, CFB at Week 4 | -0.3 (2.09)
  Carbon Dioxide, CFB at Week 8: number analyzed (Participants) | 85
  Carbon Dioxide, CFB at Week 8 | -0.6 (1.87)
  Carbon Dioxide, CFB at Week 12: number analyzed (Participants) | 86
  Carbon Dioxide, CFB at Week 12 | -0.5 (1.83)
  Chloride, Baseline (screening Week -4) | 103.7 (2.15)
  Chloride, CFB at Week 4: number analyzed (Participants) | 90
  Chloride, CFB at Week 4 | -0.3 (2.55)
  Chloride, CFB at Week 8: number analyzed (Participants) | 85
  Chloride, CFB at Week 8 | 0.6 (2.36)
  Chloride, CFB at Week 12: number analyzed (Participants) | 86
  Chloride, CFB at Week 12 | 0.5 (2.38)
  Phosphate, Baseline (screening Week -4) | 1.103 (0.1651)
  Phosphate, CFB at Week 4: number analyzed (Participants) | 90
  Phosphate, CFB at Week 4 | -0.002 (0.1836)
  Phosphate, CFB at Week 8: number analyzed (Participants) | 85
  Phosphate, CFB at Week 8 | 0.023 (0.1731)
  Phosphate, CFB at Week 12: number analyzed (Participants) | 86
  Phosphate, CFB at Week 12 | -0.015 (0.1570)

14. Secondary Outcome: Change From Baseline in Chemistry Parameter Following Administration of SC Injection: Albumin
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Grams per liter (g/L)
  Baseline (screening Week -4) | 43.1 (2.66)
  CFB at Week 4: number analyzed (Participants) | 90
  CFB at Week 4 | 0.4 (2.56)
  CFB at Week 8: number analyzed (Participants) | 85
  CFB at Week 8 | 0.8 (2.20)
  CFB at Week 12: number analyzed (Participants) | 86
  CFB at Week 12 | -0.1 (2.11)

15. Secondary Outcome: Change From Baseline in Chemistry Parameters Following Administration of SC Injection: Lipase
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Units per liter (U/L)
  Baseline (screening Week -4) | 29.4 (17.69)
  CFB at Week 4: number analyzed (Participants) | 90
  CFB at Week 4 | 0.3 (10.97)
  CFB at Week 8: number analyzed (Participants) | 85
  CFB at Week 8 | 5.6 (25.61)
  CFB at Week 12: number analyzed (Participants) | 86
  CFB at Week 12 | 1.4 (11.66)

16. Secondary Outcome: Change From Baseline in Chemistry Parameters Following Administration of SC Injection: Creatinine Clearance
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milliliter per minute (mL/min)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Milliliter per minute (mL/min)
  Baseline (screening Week -4) | 93.9 (15.15)
  CFB at Week 4: number analyzed (Participants) | 90
  CFB at Week 4 | 1.9 (6.95)
  CFB at Week 8: number analyzed (Participants) | 85
  CFB at Week 8 | 1.8 (9.37)
  CFB at Week 12: number analyzed (Participants) | 86
  CFB at Week 12 | 0.4 (8.06)

17. Secondary Outcome: Change From Baseline in Fasting Lipid Panels Following Administration of SC Injection: Total Cholesterol, High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, Triglycerides
Time Frame: Baseline (screening Week -4), and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 84
mmol/L
  Total Cholesterol, Baseline (screening Week -4) | 4.855 (0.9604)
  Total Cholesterol, CFB at Week 12: number analyzed (Participants) | 73
  Total Cholesterol, CFB at Week 12 | -0.073 (0.6056)
  HDL Cholesterol, Baseline (screening Week -4) | 1.373 (0.3764)
  HDL Cholesterol, CFB at Week 12: number analyzed (Participants) | 73
  HDL Cholesterol, CFB at Week 12 | -0.050 (0.1646)
  LDL Cholesterol, Baseline (screening Week -4) | 2.899 (0.8464)
  LDL Cholesterol, CFB at Week 12: number analyzed (Participants) | 73
  LDL Cholesterol, CFB at Week 12 | -0.040 (0.4786)
  Triglycerides, Baseline (screening Week -4) | 1.299 (0.8672)
  Triglycerides, CFB at Week 12: number analyzed (Participants) | 73
  Triglycerides, CFB at Week 12 | 0.005 (0.5692)

18. Secondary Outcome: Change From Baseline in Hematology Parameters Following Administration of SC Injection: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelet Count
Description: Blood samples were collected as assessed by protocol, at specific time points for the analysis of hematology parameters. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Giga cells per Liter (10^9 cells/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Giga cells per Liter (10^9 cells/L)
  Basophils, Baseline (screening Week -4) | 0.048 (0.0264)
  Basophils, CFB at Week 4: number analyzed (Participants) | 90
  Basophils, CFB at Week 4 | 0.000 (0.0274)
  Basophils, CFB at Week 8: number analyzed (Participants) | 85
  Basophils, CFB at Week 8 | -0.003 (0.0309)
  Basophils, CFB at Week 12: number analyzed (Participants) | 84
  Basophils, CFB at Week 12 | -0.002 (0.0343)
  Eosinophils, Baseline (screening Week -4) | 0.193 (0.1648)
  Eosinophils, CFB at Week 4: number analyzed (Participants) | 90
  Eosinophils, CFB at Week 4 | 0.006 (0.1193)
  Eosinophils, CFB at Week 8: number analyzed (Participants) | 85
  Eosinophils, CFB at Week 8 | -0.033 (0.0981)
  Eosinophils, CFB at Week 12: number analyzed (Participants) | 84
  Eosinophils, CFB at Week 12 | -0.006 (0.1198)
  Leukocytes, Baseline (screening Week -4) | 6.12 (1.901)
  Leukocytes, CFB at Week 4: number analyzed (Participants) | 90
  Leukocytes, CFB at Week 4 | 0.09 (1.524)
  Leukocytes, CFB at Week 8: number analyzed (Participants) | 85
  Leukocytes, CFB at Week 8 | -0.24 (1.364)
  Leukocytes, CFB at Week 12: number analyzed (Participants) | 84
  Leukocytes, CFB at Week 12 | -0.11 (1.210)
  Lymphocytes, Baseline (screening Week -4) | 2.076 (0.6398)
  Lymphocytes, CFB at Week 4: number analyzed (Participants) | 90
  Lymphocytes, CFB at Week 4 | 0.046 (0.4427)
  Lymphocytes, CFB at Week 8: number analyzed (Participants) | 85
  Lymphocytes, CFB at Week 8 | -0.066 (0.4864)
  Lymphocytes, CFB at Week 12: number analyzed (Participants) | 84
  Lymphocytes, CFB at Week 12 | -0.064 (0.4890)
  Monocytes, Baseline (screening Week -4) | 0.470 (0.1897)
  Monocytes, CFB at Week 4: number analyzed (Participants) | 90
  Monocytes, CFB at Week 4 | -0.006 (0.1204)
  Monocytes, CFB at Week 8: number analyzed (Participants) | 85
  Monocytes, CFB at Week 8 | -0.053 (0.1284)
  Monocytes, CFB at Week 12: number analyzed (Participants) | 84
  Monocytes, CFB at Week 12 | -0.044 (0.1448)
  Neutrophils, Baseline (screening Week -4) | 3.328 (1.3927)
  Neutrophils, CFB at Week 4: number analyzed (Participants) | 90
  Neutrophils, CFB at Week 4 | 0.054 (1.3913)
  Neutrophils, CFB at Week 8: number analyzed (Participants) | 85
  Neutrophils, CFB at Week 8 | -0.093 (1.0953)
  Neutrophils, CFB at Week 12: number analyzed (Participants) | 84
  Neutrophils, CFB at Week 12 | 0.012 (0.9941)
  Platelet Count, Baseline (screening Week -4) | 256.2 (70.85)
  Platelet Count, CFB at Week 4: number analyzed (Participants) | 89
  Platelet Count, CFB at Week 4 | -0.8 (33.28)
  Platelet Count, CFB at Week 8: number analyzed (Participants) | 85
  Platelet Count, CFB at Week 8 | -3.5 (30.93)
  Platelet Count, CFB at Week 12: number analyzed (Participants) | 83
  Platelet Count, CFB at Week 12 | 1.0 (36.35)

19. Secondary Outcome: Change From Baseline in Hematology Parameter Following Administration of SC Injection: Red Blood Cell (RBC) Count
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Trillion cells per liter (10^12/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Trillion cells per liter (10^12/L)
  Baseline (screening Week -4) | 4.74 (0.398)
  CFB at Week 4: number analyzed (Participants) | 90
  CFB at Week 4 | 0.03 (0.244)
  CFB at Week 8: number analyzed (Participants) | 85
  CFB at Week 8 | 0.01 (0.248)
  CFB at Week 12: number analyzed (Participants) | 84
  CFB at Week 12 | -0.04 (0.265)

20. Secondary Outcome: Change From Baseline in Hematology Parameter Following Administration of SC Injection: Hemoglobin
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Grams per liter (g/L)
  Baseline (screening Week -4) | 142.9 (12.14)
  CFB at Week 4: number analyzed (Participants) | 90
  CFB at Week 4 | 0.3 (7.02)
  CFB at Week 8: number analyzed (Participants) | 85
  CFB at Week 8 | -0.9 (6.87)
  CFB at Week 12: number analyzed (Participants) | 84
  CFB at Week 12 | -2.4 (7.43)

21. Secondary Outcome: Change From Baseline in Hematology Parameter Following Administration of SC Injection: Hematocrit
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood (
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Proportion of red blood cells in blood (
  Baseline (screening Week -4) | 0.4268 (0.03402)
  CFB at Week 4: number analyzed (Participants) | 90
  CFB at Week 4 | 0.0008 (0.02308)
  CFB at Week 8: number analyzed (Participants) | 85
  CFB at Week 8 | 0.0014 (0.02243)
  CFB at Week 12: number analyzed (Participants) | 84
  CFB at Week 12 | -0.0023 (0.02584)

22. Secondary Outcome: Change From Baseline in Hematology Parameter Following Administration of SC Injection: Mean Corpuscular Volume
Time Frame: Baseline (screening Week -4), Change from baseline (CFB) at Week 4, CFB at Week 8, and CFB at Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Femtoliters (fL)
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Femtoliters (fL)
  Baseline (screening Week -4) | 90.2 (4.49)
  CFB at Week 4: number analyzed (Participants) | 90
  CFB at Week 4 | -0.4 (1.74)
  CFB at Week 8: number analyzed (Participants) | 85
  CFB at Week 8 | 0.2 (2.04)
  CFB at Week 12: number analyzed (Participants) | 84
  CFB at Week 12 | 0.5 (2.51)

23. Secondary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) Less Than (<) 50 Copies Per Milliliter (c/mL) Using the Food and Drug Administration (FDA) Snapshot Algorithm - SC Injection Phase
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Percentage of participants
  Baseline (Day 1) | 100 [96 to 100]
  Week 4: number analyzed (Participants) | 91
  Week 4 | 100 [96 to 100]
  Week 8: number analyzed (Participants) | 87
  Week 8 | 99 [97 to 100]
  Week 12 | 90 [84 to 96]

24. Secondary Outcome: Percentage of Participants With Plasma HIV RNA Greater Than Equal to (>=) 50 c/mL as Per FDA Snapshot Algorithm - SC Injection Phase
Time Frame: Baseline (Day 1) and at Weeks 4, 8, 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Percentage of participants
  Baseline (Day 1) | 0 [0.0 to 3.9]
  Week 4 | 0 [0.0 to 4.0]
  Week 8: number analyzed (Participants) | 87
  Week 8 | 1.1 [0.0 to 3.4]
  Week 12 | 2.2 [0.0 to 5.1]

25. Secondary Outcome: Percentage of Participants With Protocol Defined Confirmed Virologic Failure (CVF) of >=200 c/mL - SC Injection Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. CVF was defined as rebound as indicated by two consecutive plasma HIV-1-RNA levels >=200 c/mL after prior suppression to <200 c/mL.
Time Frame: From Day 1 Up to Week 12
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Percentage of participants | 0

26. Secondary Outcome: Number of Participants With Treatment Emergent Phenotypic Resistance - SC Injection Phase
Description: Plasma samples were collected for drug resistance testing. Number of participants who met CVF criteria (two consecutive plasma HIV-1-RNA levels >=200 copies/mL after prior suppression to <200 copies/mL) with treatment emergent phenotypic resistance were reported.
Time Frame: From Day 1 Up to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Participants | 0

27. Secondary Outcome: Number of Participants With Treatment Emergent Genotypic Resistance - SC Injection Phase
Description: Plasma samples were collected for drug resistance testing. Number of participants who met CVF criteria (two consecutive plasma HIV-1-RNA levels >=200 copies/mL after prior suppression to <200 copies/mL) with treatment emergent genotypic resistance were reported.
Time Frame: From Day 1 Up to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Participants | 0

28. Secondary Outcome: Number of Participants With Post-injection Pain Assessment Using Numeric Rating Scale (NRS) on Week-3 - Screening/IM Gluteal Injection Phase
Description: A numeric rating scale was used to assess the level of pain experienced following injections with CAB + RPV. The scale contains one item and the response scale is ranging from 0= "no pain" to 10= "extreme pain". NRS questionnaire included the question regarding the maximum level of pain experienced with the most recent injections. The objective of this outcome measure was to present the data separately for each treatment received (CAB, RPV).
Time Frame: Week -3 (Baseline)
Population: Analysis was performed on sub-study safety set, which included all enrolled participants who received at least one CAB and/or RPV SC injection. The participants were analyzed according to the treatment they received. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- CAB Q4W: Participants received SC injection of CAB LA 400 mg on the left side of the body once in every 4 weeks, starting on day 1 of week 1, week 4 and week 8 during the SC abdominal injection phase and IM injections on week-4 (Screening phase), on week 12 and week 16 during Return to IM gluteal injection phase.
- RPV Q4W: Participants received SC injection of RPV LA 600 mg on the right side of the body once in every 4 weeks, starting on day 1 of week 1, week 4 and week 8 during the SC abdominal injection phase and IM injections on week-4 (Screening phase),on week 12 and week 16 during Return to IM gluteal injection phase.
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 92 | 92
Participants
  Individual item score 0 | 37 | 27
  Individual item score 1 | 21 | 16
  Individual item score 2 | 11 | 18
  Individual item score 3 | 7 | 9
  Individual item score 4 | 5 | 5
  Individual item score 5 | 1 | 6
  Individual item score 6 | 1 | 3
  Individual item score 7 | 6 | 4
  Individual item score 8 | 3 | 1
  Individual item score 9 | 0 | 1
  Individual item score 10 | 0 | 2

29. Secondary Outcome: Number of Participants With Post-injection Pain Assessment Using Numeric Rating Scale (NRS) on Week 1 - SC Injection Phase
Description: as for outcome 28
Time Frame: Day 1
Population: Analysis was performed on sub-study safety set, which included all enrolled participants who received at least one CAB and/or RPV SC injection. The participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- RPV Q4W: Participants received SC injection of RPV LA 600 mg on the right side of the body once in every 4 weeks, starting on day 1 of week 1, week 4 and week 8 during the SC abdominal injection phase and IM injections on week-4 (Screening phase), on week 12 and week 16 during Return to IM gluteal injection phase.
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 93 | 93
Participants
  Individual Item Score 0 | 16 | 22
  Individual Item Score 1 | 13 | 19
  Individual Item Score 2 | 16 | 10
  Individual Item Score 3 | 8 | 13
  Individual Item Score 4 | 6 | 2
  Individual Item Score 5 | 6 | 7
  Individual Item Score 6 | 3 | 4
  Individual Item Score 7 | 10 | 7
  Individual Item Score 8 | 6 | 5
  Individual Item Score 9 | 7 | 2
  Individual Item Score 10 | 2 | 2

30. Secondary Outcome: Number of Participants With Post-injection Pain Assessment Using NRS on Week 9- SC Injection Phase
Description: A numeric rating scale was used to assess the level of pain experienced following injections with CAB + RPV. The scale contains one item and the response scale is ranging from 0= "no pain" to 10= "extreme pain". NRS questionnaire included the questions regarding the maximum level of pain experienced with the most recent injections. The objective of this outcome measure was to present the data separately for each treatment received (CAB, RPV).
Time Frame: Week 9
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 87 | 87
Participants
  Individual Item Score 0 | 21 | 19
  Individual Item Score 1 | 9 | 11
  Individual Item Score 2 | 19 | 15
  Individual Item Score 3 | 9 | 13
  Individual Item Score 4 | 9 | 6
  Individual Item Score 5 | 4 | 7
  Individual Item Score 6 | 4 | 9
  Individual Item Score 7 | 3 | 3
  Individual Item Score 8 | 5 | 2
  Individual Item Score 9 | 4 | 0
  Individual Item Score 10 | 0 | 2

31. Secondary Outcome: Number of Participants With Post-injection Pain Assessment Using NRS on Week 13- Return to IM Gluteal Injection Phase
Description: as for outcome 30
Time Frame: Week 13
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 87 | 87
Participants
  Individual Item Score 0 | 40 | 41
  Individual Item Score 1 | 21 | 13
  Individual Item Score 2 | 10 | 12
  Individual Item Score 3 | 7 | 9
  Individual Item Score 4 | 3 | 3
  Individual Item Score 5 | 3 | 5
  Individual Item Score 6 | 0 | 2
  Individual Item Score 7 | 2 | 2
  Individual Item Score 8 | 1 | 0
  Individual Item Score 9 | 0 | 0
  Individual Item Score 10 | 0 | 0

32. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQs) Total Score -Screening/IM Gluteal Injection Phase
Description: HIVTSQ is a self-completion measure specifically designed to measure treatment satisfaction in HIV participants. HIVTSQs questionnaire includes 12 questions and the total treatment satisfaction score is computed with items 1-11 and summed to produce a total score with a possible range of 0 to 66. Higher scores indicate a greater satisfaction and a lower score indicates dissatisfaction.
Time Frame: Week -3 (Baseline)
Population: Analysis was presented only for participants in Screening/IM Gluteal Injection Phase that completed the HIVTSQs questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 93
Scores on a scale | 62.15 (5.258)

33. Secondary Outcome: HIVTSQs Total Score -SC Injection Phase
Description: as for outcome 32
Time Frame: At Week 9
Population: Analysis was presented only for participants in SC Injection Phase that completed the HIVTSQs questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 87
Scores on a scale | 51.99 (14.765)

34. Secondary Outcome: HIVTSQs Total Score -Return to IM Gluteal Injection Phase
Description: as for outcome 32
Time Frame: At Week 17
Population: Analysis was presented only for participants in Return to IM Gluteal Injection Phase that completed the HIVTSQs questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 86
Scores on a scale | 62.71 (4.217)

35. Secondary Outcome: Change From Baseline in HIVTSQs Individual Item Scores at Indicated Time Points -SC Injection Phase
Description: HIVTSQs is a 12-item questionnaire and individual item scores on HIVTSQs scale are rated as 6 (very satisfied) to 0 (very dissatisfied). Higher scores represent greater satisfaction. Data was reported for each treatment satisfaction item based on the following items: Item 1=satisfaction with current treatment, Item 2=level of HIV control based on treatment, Item 3=any side effects of present treatment, Item 4=demands made by current treatment, Item 5=convenience in finding treatment, Item 6=flexibility in finding treatment, Item 7=understanding HIV, Item 8=extent to which the treatment fits in with lifestyle, Item 9=recommendation of present treatment to someone else, Item 10=continuation with present form of treatment, Item 11=easy or difficult treatment, Item 12=amount of discomfort/pain involved with present form of treatment.
Time Frame: Baseline (Week -3) and up to Week 9
Population: Analysis was presented only for participants in SC Injection Phase that completed the HIVTSQs questionnaire. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 87
Scores on a scale
  Item 1 | -1.2 (1.85)
  Item 2 | -0.2 (0.79)
  Item 3 | -1.5 (1.93)
  Item 4 | -1.1 (1.67)
  Item 5 | -1.2 (1.88)
  Item 6 | -0.8 (1.83)
  Item 7 | -0.2 (0.93)
  Item 8 | -0.8 (1.59)
  Item 9 | -1.1 (1.68)
  Item 10 | -1.4 (1.97)
  Item 11 | -1.0 (1.47)
  Item 12 | -1.3 (1.79)

36. Secondary Outcome: Change From Baseline in HIVTSQs Individual Item Scores at Indicated Time Points - Return to IM Gluteal Injection Phase
Description: as for outcome 35
Time Frame: Baseline (Week -3) and up to Week 17
Population: Analysis was presented only for participants in Return to IM Gluteal Injection Phase that completed the HIVTSQs questionnaire. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 86
Scores on a scale
  Item 1 | 0.1 (0.43)
  Item 2 | -0.1 (0.35)
  Item 3 | 0.1 (0.72)
  Item 4 | 0.0 (0.63)
  Item 5 | 0.0 (0.55)
  Item 6 | 0.0 (0.95)
  Item 7 | 0.1 (0.55)
  Item 8 | 0.0 (0.55)
  Item 9 | 0.0 (0.32)
  Item 10 | 0.1 (0.57)
  Item 11 | 0.0 (0.58)
  Item 12 | 0.2 (0.79)

37. Secondary Outcome: Change From Study Week 9 to Study Week 17 in HIVTSQs Individual Item Scores at Indicated Time Points - Return to IM Gluteal Injection Phase
Description: as for outcome 35
Time Frame: Week 9 and Week 17
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 86
Scores on a scale
  Item 1 | 1.3 (1.77)
  Item 2 | 0.2 (0.77)
  Item 3 | 1.6 (1.85)
  Item 4 | 1.1 (1.60)
  Item 5 | 1.2 (1.78)
  Item 6 | 0.8 (1.41)
  Item 7 | 0.2 (0.83)
  Item 8 | 0.8 (1.40)
  Item 9 | 1.0 (1.68)
  Item 10 | 1.5 (1.97)
  Item 11 | 1.0 (1.39)
  Item 12 | 1.5 (1.88)

38. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Change Version (HIVTSQc) Individual Item Score at Indicated Time Points -SC Injection Phase
Description: HIVTSQc is a 12-item questionnaire to measure treatment satisfaction in HIV participants. Individual items were rated as +3 (much more satisfied) to -3(much less satisfied). Higher the score, greater the improvement in satisfaction with each aspect of treatment and lower the score, greater the deterioration in satisfaction with each aspect of treatment. Data was reported for each treatment satisfaction item based on the following items:Item 1=satisfaction with current treatment,Item2=level of HIV control based on treatment,Item3=any side effects of present treatment,Item4=demands made by current treatment,Item 5=convenience in finding treatment,Item 6=flexibility in finding treatment,Item 7=understanding HIV,Item 8=extent to which the treatment fits in with lifestyle,Item 9=recommendation of present treatment to someone else,Item 10=continuation with present form of treatment,Item 11=easy or difficult treatment,Item 12=amount of discomfort/pain involved with present form of treatment.
Time Frame: From Week -4 up to Week 9
Population: Analysis was presented only for participants in SC Injection Phase that completed the HIVTSQc questionnaire. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 87
Scores on a scale
  Item 1 | 0.7 (2.14)
  Item 2 | 1.8 (1.40)
  Item 3 | 0.5 (2.04)
  Item 4 | 1.2 (1.75)
  Item 5 | 1.0 (2.06)
  Item 6 | 1.3 (1.76)
  Item 7 | 2.0 (1.32)
  Item 8 | 1.4 (1.77)
  Item 9 | 1.3 (1.92)
  Item 10 | 0.9 (2.11)
  Item 11 | 1.2 (1.77)
  Item 12 | 0.5 (2.18)

39. Secondary Outcome: HIVTSQc Total Score at Indicated Time Points -SC Injection Phase
Description: HIVTSQ is a self-completion measure specifically designed to measure treatment satisfaction in HIV participants. Total treatment satisfaction change score is computed using items 1 to 11 and are summed to produce a score with a possible range of -33 to 33. Higher the score, greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of 0 represented no change.
Time Frame: From Week -4 up to Week 9
Population: Analysis was presented only for participants in SC Injection Phase that completed the HIVTSQc questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 87
Scores on a scale | 13.4 (17.79)

40. Secondary Outcome: Perception of Injection (PIN) Questionnaire in Domain Scores and Individual Item Scores- Screening/IM Gluteal Injection Phase
Description: The PIN questionnaire is characterized by the dimension scores based on 4 domains including Bother from injection site reactions (ISRs), Acceptability, Leg movement and Sleep categories. The objective of this endpoint is to present analysis of 2 (out of 4) PIN domains: Bother from ISRs and Acceptability. This questionnaire contains 21 items that measure pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside of a clinical trial. Domain scores were calculated as a mean of all items with the domain. Scores range from 1 to 5,and questions are phrased in such a way as to ensure that 1 always equated with the most favorable perception of vaccination, and 5 the most unfavorable. Higher scores represent worse perception of injection. The objective of this outcome measure was to present the data separately for each treatment received (CAB, RPV).
Time Frame: At Week -3 (Baseline)
Population: Analysis was presented only for participants in Screening/IM Gluteal Injection Phase that completed the PIN questionnaire based on intervention received. The participants were analyzed according to the treatment they received.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 93 | 93
Scores on a scale
  Bother of ISRs | 1.44 (0.484) | 1.53 (0.568)
  Acceptance | 1.51 (0.676) | 1.71 (0.781)

41. Secondary Outcome: PIN Questionnaire in Domain Scores and Individual Item Scores at Indicated Time Points - SC Injection Phase
Description: as for outcome 40
Time Frame: At Week 1 and Week 9
Population: Analysis was presented only for participants in SC Injection Phase that completed the PIN questionnaire based on intervention received. The participants were analyzed according to the treatment they received. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 93 | 93
Scores on a scale
  Bother of ISRs, Week 1 | 2.23 (0.918) | 1.95 (0.913)
  Bother of ISRs, Week 9: number analyzed (Participants) | 87 | 87
  Bother of ISRs, Week 9 | 2.10 (0.964) | 1.93 (0.891)
  Acceptance, Week 1 | 2.60 (1.173) | 2.28 (1.167)
  Acceptance, Week 9: number analyzed (Participants) | 87 | 87
  Acceptance, Week 9 | 2.30 (1.206) | 2.12 (1.156)

42. Secondary Outcome: PIN Questionnaire in Domain Scores and Individual Item Scores - Return to IM Gluteal Injection Phase
Description: as for outcome 40
Time Frame: At Week 13
Population: Analysis was presented only for participants in Return to IM Gluteal Injection Phase that completed the PIN questionnaire based on intervention received. The participants were analyzed according to the treatment they received. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 87 | 87
Scores on a scale
  Bother of ISRs | 1.23 (0.358) | 1.28 (0.377)
  Acceptance | 1.32 (0.570) | 1.46 (0.679)

43. Secondary Outcome: Change From Baseline to the PIN Questionnaire in Domain Scores and Individual Item Scores at Indicated Time Points - SC Injection Phase
Description: as for outcome 40
Time Frame: Change from Baseline (Week -3) at Week 1 and Week 9
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 93 | 93
Scores on a scale
  Bother of ISRs, Change from Baseline at Week 1 | 0.79 (0.843) | 0.41 (0.909)
  Bother of ISRs, Change from Baseline at Week 9: number analyzed (Participants) | 87 | 87
  Bother of ISRs, Change from Baseline at Week 9 | 0.70 (0.931) | 0.41 (0.877)
  Acceptance, Change from Baseline at Week 1 | 1.09 (1.100) | 0.58 (1.177)
  Acceptance, Change from Baseline at Week 9: number analyzed (Participants) | 87 | 87
  Acceptance, Change from Baseline at Week 9 | 0.86 (1.145) | 0.44 (1.103)

44. Secondary Outcome: Change From Baseline to the PIN Questionnaire in Domain Scores and Individual Item Scores at Indicated Time Points - Return to IM Gluteal Injection Phase
Description: as for outcome 40
Time Frame: Change from Baseline (Week -3) at Week 13
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB Q4W | RPV Q4W
Number analyzed (Participants) | 87 | 87
Scores on a scale
  Bother of ISRs | -0.17 (0.369) | -0.24 (0.537)
  Acceptance | -0.12 (0.719) | -0.22 (0.888)

45. Secondary Outcome: Number of Participants With Their Treatment Preference Assessed Using Preference Questionnaire on Week 9 - SC Injection Phase
Description: A preference questionnaire was used to assess participant's preference for the subcutaneous injections compared with the gluteal injections. The "Preference" questionnaire included a single item question evaluating preference of HIV treatment. Participants were required to provide their response to Question, which stated "Which injection site do you prefer". The responses included Intramuscular Injections in the buttock, Subcutaneous Injections in the Abdomen and No preference.
Time Frame: Up to Week 9
Population: Analysis was presented only for participants in SC Injection Phase that completed the Preference questionnaire. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 85
Participants
  Intramuscular Injections in the buttock | 50
  Subcutaneous Injections in the Abdomen | 29
  No preference | 6

46. Secondary Outcome: Number of Participants With Their Treatment Preference Assessed Using Preference Questionnaire on Week 17 - Return to IM Gluteal Injection Phase
Description: as for outcome 45
Time Frame: Up to Week 17
Population: Analysis was presented only for participants in Return to IM Gluteal Injection Phase that completed the Preference questionnaire. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabotegravir Long Acting (CAB LA) 400 Milligrams (mg) + Rilpivirine Long Acting (RPV) LA 600 mg
Number analyzed (Participants) | 87
Participants
  Intramuscular Injections in the buttock | 61
  Subcutaneous Injections in the Abdomen | 21
  No preference | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected from Week -4 for screening/Gluteal injection phase, from day 1 up to 12 weeks for SC Injection Phase and from Week 12 to Week 20 for Return to IM Gluteal Injection Phase.
Description: All-cause mortality, Non-SAEs and SAEs were reported based on the sub-study Enrolled population for the CAB LA 400 mg + RPV LA 600 mg -Screening Phase group, and based on Safety population for CAB LA 400 mg +RPV LA 600 mg - SC Injection Phase and CAB LA 400 mg +RPV LA 600 mg -Return to IM Gluteal Injection Phase groups. AEs were presented phase-wise.
Groups:
- CAB LA 400 mg + RPV LA 600 mg - Screening Phase: Participants received a single IM gluteal injection of CAB LA 400 mg and RPV LA 600 mg prior to the administration of SC injection on Week -4 during the Screening Phase.
- CAB LA 400 mg + RPV LA 600 mg - SC Injection Phase: Participants received a SC injection of CAB LA 400 mg and RPV LA 600 mg on Day 1 in every 4 weeks (Q4W) for a total of 12 weeks during the SC abdominal Injection Phase.
- CAB LA 400 mg + RPV LA 600 mg - Return to IM Gluteal Injection Phase: Participants received first IM gluteal injection (at Week 12 and week 16) of CAB LA 400 mg + RPV LA 600 mg during the return to Gluteal Injection Phase and subsequent gluteal injection occurred after Q4W.
Arm/Group | CAB LA 400 mg + RPV LA 600 mg - Screening Phase | CAB LA 400 mg + RPV LA 600 mg - SC Injection Phase | CAB LA 400 mg + RPV LA 600 mg - Return to IM Gluteal Injection Phase
All-Cause Mortality (participants affected / at risk) | 1/94 | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/93 | 0/93
Other Adverse Events (participants affected / at risk) | 33/94 | 85/93 | 38/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA 400 mg + RPV LA 600 mg - Screening Phase (N=94) | CAB LA 400 mg + RPV LA 600 mg - SC Injection Phase (N=93) | CAB LA 400 mg + RPV LA 600 mg - Return to IM Gluteal Injection Phase (N=93)
Passed away due to unknown reasons (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA 400 mg + RPV LA 600 mg - Screening Phase (N=94) | CAB LA 400 mg + RPV LA 600 mg - SC Injection Phase (N=93) | CAB LA 400 mg + RPV LA 600 mg - Return to IM Gluteal Injection Phase (N=93)
Injection site pain (General disorders) | 29 (55) | 69 (260) | 30 (59)
Injection site nodule (General disorders) | 3 (4) | 60 (183) | 9 (13)
Injection site erythema (General disorders) | 0 (0) | 48 (142) | 1 (2)
Injection site swelling (General disorders) | 0 (0) | 29 (66) | 1 (2)
Injection site induration (General disorders) | 0 (0) | 24 (66) | 2 (3)
Injection site pruritus (General disorders) | 2 (2) | 19 (40) | 1 (2)
Injection site warmth (General disorders) | 0 (0) | 11 (22) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 7 (12) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 6 (8) | 1 (1)
Injection site discolouration (General disorders) | 0 (0) | 6 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT05896748/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05896748/SAP_001.pdf